CLINICAL TRIAL: NCT02906293
Title: AbStats: Assessing Post-Prandial Intestinal Event Rates in Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Almario, Health Services Research Scientist, Cedars-Sinai Medical Center
Other Study IDs: Pro00045465
Record Dates: First submitted 2016-09-07; First posted 2016-09-20 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Post-prandial Intestinal Rates

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Participants: Potential participants will self-refer.
  Interventions: Other: Abdominal acoustic measurement

INTERVENTIONS:
Other: Abdominal acoustic measurement — On Day 1 participants will record their intestinal rate at baseline fasting, pre-"small meal," and upon completion of the meal. On Day 2 participants will record their intestinal rate at baseline fasting, pre-"large meal," and upon completion of meal.

SUMMARY:
This study seeks to: Assess "normal" intestinal event rates for healthy subjects, to determine the effect of meal size on an individual's intestinal rate, and to determine whether there are differences between individuals in the fasting and post-prandial setting.

The investigators hypothesize the following:

1. Fasting intestinal rate will be consistently less than 14 events per minute, similar to previously documented bowel sound frequency.
2. There will a uniform increase in intestinal rate in the immediate post-prandial setting. There will be direct correlation between maximal and average post-prandial intestinal rates and meal size. Likewise, meal size will correlate with time to baseline fasting intestinal rate.
3. Males and those with lower body mass index (BMI) will experience higher maximal and average post-prandial intestinal rates and shorter time to baseline fasting levels compared to females and those with higher BMI, respectively.

DETAILED DESCRIPTION:
Participants will complete a baseline demographic and medical data sheet comprising of age, gender, race, ethnicity, height, weight, education, employment status, past medical history, and current prescription and over-the-counter medications. An AbStats device along with a log sheet will be provided to each subject, both of which will be returned upon completion of participation.

Upon waking, prior to oral intake, participants will place the AbStats disposable sensor on their abdomen and secure it using adhesive tape. The sensor is connected to a monitor which records the sounds collected by the sensors and interprets them to create and intestinal rate reading, measured as acoustic events per minute. The device will display a numerical intestinal rate reading, measured as acoustic events per minute. The device will display a numerical intestinal rate that participants will record on their personal log sheet. The purpose of this value is to assess the intestinal rate during fasting.

Participants will then eat a small standardized breakfast comprised of a thinkThin oatmeal single serve bowl, toasted English muffin with butter, and an 11oz iced coffee. No additions or substitutions are permitted in order to standardize the meal. The percent of food eaten will be recorded on the log sheet.

Lunch on Day 1 will be a "small meal" consisting of half of a turkey and Swiss Corner Bakery sandwich, cup of fruit, and 12oz can of diet soda. It will be eaten four to five hours after breakfast. No snacks are permitted between breakfast and lunch. Again, a pre-meal intestinal rate reading will be obtained 30 minutes prior to eating lunch; participants will secure the device onto the abdomen multiple times in order to gather post-prandial data. The intestinal rate will be recorded on the log sheet. The subject will record intestinal rate every 30 minutes for 5 hours after completion of the meal (e.g., lunch at 12 pm, then place sensors on abdomen for 10 minutes at 12:30 pm, 1:00 pm, 1:30 pm, 2:00 pm, 2:30 pm, 3:00 pm, 3:30 pm, 4: 00 pm, 4:30 pm, and 5:00 pm). Afterwards, participants can eat freely once these data points have been obtained. Dinner will be a meal of their choosing.

Day 2 of the study will be largely similar to Day 1: participants will measure fasting intestinal rate upon waking and will eat a standardized breakfast (see above). The main difference in Day 2 is that participants will eat a "large meal" for lunch consisting of a full turkey and Swiss Corner Bakery sandwich, cup of fruit, small bag of potato chips, small cookie, and a 12oz can of diet soda. The same pre- and post-lunch measurements notes above will be measured and recorded. By performing the above, investigators will assess preliminary intestinal rate measurements in the fasting state, after a small lunch (Day 1), and after a large lunch (Day 2).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 65 years
* Able to provide consent

Exclusion Criteria:

* Age younger than 18 or older than 65 years
* Unable to provide consent
* Vegetarian or vegan
* Pregnant
* Prior intestinal surgery
* Recent gastroenteritis, diverticulitis or stool infection within past 3 months
* Diagnosis of irritable bowel syndrome
* Diagnosis of inflammatory bowel disorder (Crohn's disease, ulcerative colitis, indeterminate colitis, microscopic colitis, gastritis or enterocolitis).
* Diagnosis of a malabsorption disorder: Celiac disease, protein losing enteropathy, pancreatic insufficiency, etc.
* Diagnosis of autoimmune disorder: diabetes mellitus, scleroderma, undifferentiated connective tissue disorder, etc.
* Diagnosis of motility disorder: achalasia, esophageal spasm, outlet obstruction, gastroparesis, chronic constipation, etc.
* History of acute pancreatitis within past 3 months
* History of GI malignancy (stomach, small or large intestine, pancreatic, neuroendocrine tumor, etc.)
* Current or recent treatment with chemotherapy within past 3 months
* History of radiation treatment
* Current or recent use (within past month) of medications that either promote or decrease motility: opioids, cholinergic agonists, opioid antagonists, anti-diarrheals, pro-kinetic medications (e.g., metoclopramide, domperidone, erythromycin), etc.
* Antibiotic use within 3 months
* Diabetes mellitus with HgA1C >6.0

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Baseline fasting intestinal rate | 10 minutes
  Prior to any oral intake, participants will record intestinal rate for 10 minutes
Pre-meal intestinal rate | 30 minutes prior to eating lunch participants will secure the device and record for 10 minutes
Post-prandial intestinal rate | Every 30 minutes for 5 hours after completion of meal

CONTACTS AND LOCATIONS:
Overall Officials: Christopher V. Almario, MD, MSHPM, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baid H. A critical review of auscultating bowel sounds. Br J Nurs. 2009 Oct 8-21;18(18):1125-9. doi: 10.12968/bjon.2009.18.18.44555. PMID 19966732
- [Background] Felder S, Margel D, Murrell Z, Fleshner P. Usefulness of bowel sound auscultation: a prospective evaluation. J Surg Educ. 2014 Sep-Oct;71(5):768-73. doi: 10.1016/j.jsurg.2014.02.003. Epub 2014 Apr 24. PMID 24776861
- [Background] Spiegel BM, Kaneshiro M, Russell MM, Lin A, Patel A, Tashjian VC, Zegarski V, Singh D, Cohen SE, Reid MW, Whitman CB, Talley J, Martinez BM, Kaiser W. Validation of an acoustic gastrointestinal surveillance biosensor for postoperative ileus. J Gastrointest Surg. 2014 Oct;18(10):1795-803. doi: 10.1007/s11605-014-2597-y. Epub 2014 Aug 5. PMID 25091837
- [Background] Kaneshiro M, Kaiser W, Pourmorady J, Fleshner P, Russell M, Zaghiyan K, Lin A, Martinez B, Patel A, Nguyen A, Singh D, Zegarski V, Reid M, Dailey F, Xu J, Robbins K, Spiegel B. Postoperative Gastrointestinal Telemetry with an Acoustic Biosensor Predicts Ileus vs. Uneventful GI Recovery. J Gastrointest Surg. 2016 Jan;20(1):132-9; discussion 139. doi: 10.1007/s11605-015-2956-3. Epub 2015 Sep 25. PMID 26408329